CLINICAL TRIAL: NCT06677177
Title: The Efficacy of Nano-water in Combination With Tamsulosin-Dutasteride for Alleviating Lower Urinary Tract Symptoms in Men With Benign Prostatic Hyperplasia
Brief Title: The Efficacy of Nano-water in Combination With Tamsulosin- Dutasteride for Lower Urinary Tract Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALI KAMAL M. SAMI (Other)
Collaborators: University of Sulaimani (Other)
Responsible Party: Sponsor-Investigator, ALI KAMAL M. SAMI, Lecturer , Urology , Department of Surgery, College of Medicine, Medical Doctor, University of Sulaimani
Organization: University of Sulaimani (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 574
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower urinary tract symptoms; benign Prostate Hyperplasia; Tamsulosin; Dutasteride; Nano-water; International Prostate Symptom Score IPSS
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Tamsulosin; Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with LUTS due to BPH/ nano-water (Experimental): Patients with Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia receiving nano-water combined with tamsulosin and Dutasteride
  Interventions: Dietary Supplement: Nano-water, Tamsulosin Dutasteride
- Patients with LUTS due to BPH/regular water (Active Comparator): Patients with Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia receiving regular water combined with tamsulosin and Dutasteride
  Interventions: Drug: Regular water, tamsulosin, Dutasteride

INTERVENTIONS:
Dietary Supplement: Nano-water, Tamsulosin Dutasteride — Nano-water, given in a dose of 20 ml/kg daily for a period of 3 months Tamsulosin capsule in a dose of 0.4mg daily for a period of 3 months Dutasteride tablet in a dose of 0.5mg daily for a period of 3 months
  Other Names: Tamsulosin; Dutasteride
  Arms: Patients with LUTS due to BPH/ nano-water
Drug: Regular water, tamsulosin, Dutasteride — Regular water, given in a dose of 20 ml/kg daily for a period of 3 months Tamsulosin capsule in a dose of 0.4mg daily for a period of 3 months Dutasteride tablet in a dose of 0.5mg daily for a period of 3 months
  Other Names: Tamsulosin; Dutasteride
  Arms: Patients with LUTS due to BPH/regular water

SUMMARY:
The goal of this clinical trial is to learn if nano-water combined with tamsulosin and dutasteride can relieve the symptoms of lower urinary tract symptoms in adults with benign prostatic hyperplasia . The main questions it aims to answer are:

Does nano-water improve the results of treating patients with lower urinary tract symptoms? What is the difference between the medications alone and the medications with nano-water? Researchers will compare nano-water to a placebo (an ordinary bottled drinking water) to see if nano-water works to treat lower urinary tract symptoms .

Participants will:

Take (nano-water combined with Tamsulosin and Dutasteride) or a placebo an (ordinary bottled drinking water) combined with Tamsulosin and Dutasteride every day for 3 months Visit the clinic once every 4 weeks for checkups Keep a diary of their symptoms and the frequency of these symptoms

DETAILED DESCRIPTION:
Introduction Symptoms of lower urinary tract (LUT) are the most prevalent complaint among men diagnosed with benign prostatic hyperplasia (BPH). Men who have symptoms of LUT because of BPH (LUT/BPH) are more likely to seek medical attention when their symptoms become unbearable. The symptoms of LUT/BPH are usually related to voiding or storage. It has been discovered that the frequency of symptoms of LUT rises in a linear manner with age. Alpha-blockers and five alpha-reductase inhibitors have been combined to treat males with symptoms of LUT due to BPH conservatively. Structured water, a nanotechnology product, possesses unique qualities that set it apart from conventional water. Subjecting water to electromagnetic and other energy fields created and imbued it with its distinct properties.

Water that has had its molecules altered to form smaller clusters of water molecules is known as Nano-water. Conventional water comprises larger clusters of water molecules (H2O) joined by hydrogen bonds. In Nano-water, these clusters are smaller and usually comprise smaller-than-normal water structures like hexagonal or tetrahedral formations. More compact water clusters and a decrease in the propensity of water molecules to the group, often creating smaller, more stable structures-also enhanced-are the unique Nano-water components. Hydrogen Bonding: Changes to the hydrogen bonding network give the water additional structure.

Finally, improved Solubility: Minerals and other substances are more soluble due to the altered molecular arrangement. Nanotechnology, engineering, and manipulation of materials at the nanoscale (1-100 nm) provide Nano-water's potential. With this method, researchers can study and experiment with water-based nano-materials. Nano-water's unique structure is thought to improve water quality, which could have several health advantages. Among these is increased hydration due to Nano-water's smaller molecular clusters' easier passage through cell membranes, improving waste removal and nutrient transport efficiency. Studies indicate that compared to other substances, Nano-water may have a more significant potential for antioxidants. Some of its benefits are effectively combating harmful free radicals, reducing oxidative stress, and possibly reducing the risk of inflammation and chronic illnesses. Additionally, Nano-water may improve detoxification and support healthy kidney and liver function by more efficiently binding to toxins and heavy metals. It shows it induces better Circulation: Because Nano-water is said to have a lower viscosity, blood flow may be enhanced, resulting in more effective delivery of nutrients and oxygen to tissues and organs.

Water structured by nanotechnology: Magnalife is produced by modulators., particular energy fields, and frequencies that change regular water into Nano-water.

The study aimed to assess the effectiveness of Nano-water doubled with tamsulosin-dutasteride in improving symptoms of LUT in BPH patients.

Patients and methods From February 2016 to November 2022, a double-blind, randomized study was carried out in Sulaimani, Iraq, in the Kurdistan region.

A questionnaire determined our patients' International Prostatic Symptom Score (IPSS). Peak urine low rates (Qmax) were calculated, and residual urine (RU) was evaluated along with an ultrasound examination of the prostate's size.

The study excluded all patients with high prostatic-specific antigens and urinary tract infections. Two groups comprising 210 men were randomly assigned for three months based on their prostate volume (>30 and < 80 ccs) and an IPSS ≥ 13 or higher. Two groups of one hundred and five men each were given different amounts of the medication: group A received Nano-water with tamsulosin-dutasteride. In contrast, Group B was given regular water with the same medication.

Unlabeled water was given in a daily dosage of 20 milliliters per kilogram of body weight-with tamsulosin 0.4 mg and finasteride 0.5 mg. At the start (baseline data) and the end of the three months, both groups underwent evaluations for the IPSS, Qmax, and RU.

The Ethics Committee of the University of Sulaimani College of Medicine authorized the current study. All individuals provided informed consent.

The statistical analysis for the study was carried out using SPSS version 24. The data were coded, tallied, and presented descriptively. Inferential data techniques, including descriptive statistics like frequency, percentage, mean, standard deviation, and the Chi-squared test, were used in the analysis. The significance of the test results was assessed using probabilistic criteria based on P-value. Specifically, a P-value of 0.05 or higher was regarded as non-significant, less than 0.001 as highly significant, and less than 0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* prostate size >30 cc and < 80 cc
* IPSS >13

Exclusion Criteria:

* High serum PSA
* Urinary tract infections

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with benign prostatic hyperplasia
Enrollment: 210 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptoms Score IPSS | From enrollment to the end of treatment at 3 months
  International Prostate Symptoms Score IPSS include 7 questions , to which each question is given a number of 1-5 , these questions include:
  Frequency, Urgency, Hesitancy, Nocturia, Incomplete emptying, Weak stream, Straining.
Qmax | From enrollment to the end of treatment at 3 months
  Qmax is the maximum flow rate of urine measure by a Flowmetry device and expressed in ml/second
Residual Urine | From enrollment to the end of treatment at 3 months
  Residual Urine is the post-voiding residual volume of urine remaining in the urinary bladder after voiding, measure by an ultrasound machine and expressed in ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ali K M. Sami, Principal Investigator — College of Medicine, University of Sulaimani
Locations (1):
- College of Medicine, Sulaymaniyah, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
Because of the social traditions here that patients do not want their private details and personal informations to be shared to other non treating doctors and they agreed to participate in this clinical trials being confirmed that the confidentiality of their personal details will not be shared.